CLINICAL TRIAL: NCT06003829
Title: A RANDOMIZED, PHASE 1, SINGLE-BLIND, MULTI-PERIOD STUDY TO INVESTIGATE THE PALATABILITY OF PF-07923568 ORAL SUSPENSION IN DIFFERENT LIQUID VEHICLES IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn About the Tastes of Different Suspensions With the Study Medicine (PF-07923568) in Healthy Adult Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: C5241014; 2023-504924-24-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-07-26; First posted 2023-08-22 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — denatonium

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental)
  Interventions: Drug: Sinsunatovir
- Treatment B (Experimental)
  Interventions: Drug: Sinsunatovir
- Treatment C (Other): Comparator
  Interventions: Other: Bitrex
- Treatment D (Experimental)
  Interventions: Drug: Sinsunatovir
- Treatment E (Experimental)
  Interventions: Drug: Sinsunatovir
- Treatment F (Experimental)
  Interventions: Drug: Sinsunatovir

INTERVENTIONS:
Drug: Sinsunatovir — Single dose, to be spit out after tasting
  Arms: Treatment A; Treatment B; Treatment D; Treatment E; Treatment F
Other: Bitrex — Single dose, to be spit out after tasting
  Arms: Treatment C

SUMMARY:
The purpose of this study is to learn about the tastes of different suspensions with the study medicine called PF-07923568 in healthy adult participants. In a suspension, the medicine is mixed with a liquid, usually water, in which it cannot dissolve and therefore remains intact in the form of small particles.

This study is seeking for healthy participants who:

* are aged 18 years of age or older.
* can produce a baby must agree to use a highly effective method of birth control.
* are confirmed to be healthy by some medical tests. This study can include both men and women.
* have body mass index (BMI) of 16 to 32 kg/m2 and a total body weight of more than 45 kilograms.

Participants will take sisunatovir prepared in 5 different suspensions and bitrex over two days to see if they are good to taste. Participants will answer a questionnaire after tasting each suspension. The questionnaire will be completed for each suspension. The questionnaire asks participants to test each suspension at 4 different times after tasting and spitting out the suspension. At least 60 minutes will pass between tasting each suspension.

The total planned time period of participation is around 5 to 8 weeks. This includes the screening period of up to 28 days. Followed by first administration of study medicine. Then a 3 day in-patient stay at the study clinic. It also includes a follow-up phone call that happens 28-35 days after the final taste test.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, blood pressure, pulse rate and standard 12-lead electrocardiogram (ECG).
* Body mass index (BMI) of 16-32 kg/m2; and a total body weight >45 kg

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine,pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Conditions that affect ability to taste eg, dysgeusia, respiratory infection, cold, etc.
* History of hypersensitivity to the active compounds or to any inactive ingredients (excipients) contained in the formulations.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
* A positive urine drug test at screening or admission.
* A positive serum pregnancy test at screening and/or positive urine/serum pregnancy test in woman/women of childbearing potential (WOCBP) at Day -1
* Use of tobacco/nicotine containing products
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm Hg for participants ≥60 years old, following at least 5 minutes of supine rest.
* Renal impairment as defined by an estimated glomerular filtration rate (eGFR) (units of mL/min/1.73m²) <60 mL/min(/1.73m²) based on 2021 chronic kidney disease epidemiology (CKD-EPI).
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin (Bili) ≥ 1.05 × upper limit of normal (ULN). Participants with an elevated total bilirubin consistent with Gilbert's Disease should have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants were enrolled in the study.
Pre-assignment Details: Participants received sisunatovir prepared in 5 different suspensions (formulation A, B, D, E and F) and bitrex (formulation C as comparator).
Groups:
- Formulation A Then B Then D Then C Then A Then E Then None Then F: Participants were randomized to receive formulation A then B then D and then C in Period 1, 2, 3 and 4 respectively, on Day 1 of the study. On Day 2 of the study participants received formulation A then E then no formulation and then formulation F in Period 5, 6, 7 and 8 respectively. A single dose of each formulation was administered. There was at least 60 minutes interval between each study formulation.
- Formulation B Then C Then A Then D Then E Then F Then A Then None: Participants were randomized to receive formulation B then C then A and then D in Period 1, 2, 3 and 4 respectively, on Day 1 of the study. On Day 2 of the study participants received formulation E then F then A and then no formulation in Period 5, 6, 7 and 8 respectively. A single dose of each formulation was administered. There was at least 60 minutes interval between each study formulation.
- Formulation C Then D Then B Then A Then F Then None Then E Then A: Participants were randomized to receive formulation C then D then B and then A in Period 1, 2, 3 and 4 respectively, on Day 1 of the study. On Day 2 of the study participants received formulation F then None then E and then A in Period 5, 6, 7 and 8 respectively. A single dose of each formulation was administered. There was at least 60 minutes interval between each study formulation.
- Formulation D Then A Then C Then B Then None Then A Then F Then E: Participants were randomized to receive formulation D then A then C then B in Period 1, 2, 3 and 4 respectively, on Day 1 of the study. On Day 2 of the study participants received no formulation then formulation A then F then E in Period 5, 6, 7 and 8 respectively. A single dose of each formulation was administered. There was at least 60 minutes interval between each study formulation.
Period: Period 1 (Day 1 of the Study)
Arm/Group | Formulation A Then B Then D Then C Then A Then E Then None Then F | Formulation B Then C Then A Then D Then E Then F Then A Then None | Formulation C Then D Then B Then A Then F Then None Then E Then A | Formulation D Then A Then C Then B Then None Then A Then F Then E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 (Day 1 of the Study)
Arm/Group | Formulation A Then B Then D Then C Then A Then E Then None Then F | Formulation B Then C Then A Then D Then E Then F Then A Then None | Formulation C Then D Then B Then A Then F Then None Then E Then A | Formulation D Then A Then C Then B Then None Then A Then F Then E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 3 (Day 1 of the Study)
Arm/Group | Formulation A Then B Then D Then C Then A Then E Then None Then F | Formulation B Then C Then A Then D Then E Then F Then A Then None | Formulation C Then D Then B Then A Then F Then None Then E Then A | Formulation D Then A Then C Then B Then None Then A Then F Then E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 4 (Day 1 of the Study)
Arm/Group | Formulation A Then B Then D Then C Then A Then E Then None Then F | Formulation B Then C Then A Then D Then E Then F Then A Then None | Formulation C Then D Then B Then A Then F Then None Then E Then A | Formulation D Then A Then C Then B Then None Then A Then F Then E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 5 (Day 2 of the Study)
Arm/Group | Formulation A Then B Then D Then C Then A Then E Then None Then F | Formulation B Then C Then A Then D Then E Then F Then A Then None | Formulation C Then D Then B Then A Then F Then None Then E Then A | Formulation D Then A Then C Then B Then None Then A Then F Then E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 6 (Day 2 of the Study)
Arm/Group | Formulation A Then B Then D Then C Then A Then E Then None Then F | Formulation B Then C Then A Then D Then E Then F Then A Then None | Formulation C Then D Then B Then A Then F Then None Then E Then A | Formulation D Then A Then C Then B Then None Then A Then F Then E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 7 (Day 2 of the Study)
Arm/Group | Formulation A Then B Then D Then C Then A Then E Then None Then F | Formulation B Then C Then A Then D Then E Then F Then A Then None | Formulation C Then D Then B Then A Then F Then None Then E Then A | Formulation D Then A Then C Then B Then None Then A Then F Then E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 8 (Day 2 of the Study)
Arm/Group | Formulation A Then B Then D Then C Then A Then E Then None Then F | Formulation B Then C Then A Then D Then E Then F Then A Then None | Formulation C Then D Then B Then A Then F Then None Then E Then A | Formulation D Then A Then C Then B Then None Then A Then F Then E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled analysis set included participants if the informed consent was not withdrawn prior to participating in any study activity after screening.
Groups:
- All Participants: All participants who were enrolled and received study intervention in a randomized crossover manner at each period, up to 4 times a day on Day 1 or Day 2.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.00 (18.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Sensory Attributes Based on Palatability Assessment Questionnaire at 1 Minute Post-dose on Day 1
Description: Participants were offered formulation for tasting where they had to swirl sample in their mouth for approximately 10 seconds, and then spit it out. Participant had to assess each sensory attribute on scale of 0 (good) to 100 (bad) after tasting formulation, lower score= better palatability. Following were sensory attributes: mouth feel (grittiness/stickiness or waxiness, 0= normal mouth feel,100=bad mouth feel);bitterness (degree of bitterness of the product, 0= not bitter at all,100= extremely bitter); sweetness(degree of sweet taste,0=sweet, 100= not sweet at all); sourness (degree of sour taste,0= not sour at all,100= extremely sour);saltiness(degree of salty taste,0=not salty at all,100= extremely salty); tongue/mouth burn(degree of tongue/mouth burn,0= no burn at all,100= extreme burn);overall liking (how much like or dislike product, 0= like, 100= dislike).Mean score for each sensory attributes based on palatability assessment questionnaire are reported in this outcome measure.
Time Frame: At 1 minute after tasting specified study formulation on Day 1
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Data was reported only for those formulations which were administered on Day 1.
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Groups:
- Formulation A: Participants received single dose of formulation A of sisunatovir. Participants had to swirl the formulation in the mouth for approximately 10 seconds, and then spit it out.
- Formulation B: Participants received single dose of formulation B of sisunatovir. Participants had to swirl the formulation in the mouth for approximately 10 seconds, and then spit it out.
- Formulation C: Participants received single dose of bitrex. Participants had to swirl the formulation in the mouth for approximately 10 seconds, and then spit it out.
- Formulation D: Participants received single dose of formulation D of sisunatovir. Participants had to swirl the formulation in the mouth for approximately 10 seconds, and then spit it out.
Arm/Group | Formulation A | Formulation B | Formulation C | Formulation D
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale
  Mouth Feel | 80.3 [72.65 to 88.02] | 49.4 [40.69 to 58.15] | 54.0 [40.09 to 67.91] | 48.5 [37.47 to 59.53]
  Bitterness | 80.2 [73.91 to 86.43] | 49.8 [36.55 to 62.95] | 59.5 [47.10 to 71.90] | 49.4 [34.47 to 64.36]
  Sweetness | 25.8 [8.89 to 42.61] | 36.3 [26.57 to 45.93] | 16.3 [7.46 to 25.04] | 28.3 [16.59 to 40.08]
  Sourness | 50.1 [35.25 to 64.92] | 32.8 [23.49 to 42.18] | 32.8 [16.65 to 49.01] | 30.3 [17.85 to 42.82]
  Saltiness | 46.6 [30.18 to 62.99] | 28.0 [17.18 to 38.82] | 26.1 [13.18 to 38.99] | 30.8 [18.46 to 43.20]
  Tongue/Mouth Burn | 27.5 [13.30 to 41.70] | 21.3 [10.72 to 31.78] | 14.8 [6.03 to 23.63] | 18.3 [8.50 to 28.17]
  Overall Liking | 85.1 [76.58 to 93.59] | 55.6 [43.51 to 67.65] | 57.9 [45.23 to 70.60] | 50.4 [36.49 to 64.35]

2. Primary Outcome: Mean Score of Sensory Attributes Based on Palatability Assessment Questionnaire at 5 Minutes Post-dose on Day 1
Description: as for outcome 1
Time Frame: At 5 minutes after tasting specified study formulation on Day 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Formulation A | Formulation B | Formulation C | Formulation D
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale
  Mouth Feel | 66.6 [56.85 to 76.31] | 45.8 [33.91 to 57.59] | 50.9 [39.47 to 62.36] | 46.7 [32.36 to 60.97]
  Bitterness | 72.3 [61.87 to 82.63] | 45.9 [37.18 to 54.66] | 53.5 [42.36 to 64.64] | 53.2 [40.82 to 65.52]
  Sweetness | 22.7 [9.28 to 36.05] | 30.3 [18.94 to 41.56] | 18.3 [8.72 to 27.95] | 27.4 [14.88 to 39.95]
  Sourness | 43.8 [28.95 to 58.71] | 30.3 [20.83 to 39.83] | 28.9 [15.76 to 42.08] | 27.7 [17.09 to 38.24]
  Saltiness | 34.5 [18.43 to 50.57] | 23.0 [13.24 to 32.76] | 24.9 [12.22 to 37.61] | 24.5 [12.84 to 36.16]
  Tongue/Mouth Burn | 23.3 [10.50 to 36.16] | 21.8 [11.07 to 32.60] | 17.1 [7.42 to 26.75] | 17.3 [7.37 to 27.13]
  Overall Liking | 78.3 [68.19 to 88.31] | 53.3 [38.59 to 68.07] | 52.3 [40.97 to 63.70] | 49.4 [34.27 to 64.56]

3. Primary Outcome: Mean Score of Sensory Attributes Based on Palatability Assessment Questionnaire at 10 Minutes Post-dose on Day 1
Description: as for outcome 1
Time Frame: At 10 minutes after tasting specified study formulation on Day 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Formulation A | Formulation B | Formulation C | Formulation D
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale
  Mouth Feel | 62.6 [50.44 to 74.72] | 43.2 [31.29 to 55.04] | 40.3 [32.23 to 48.27] | 44.6 [29.45 to 59.71]
  Bitterness | 66.2 [52.84 to 79.49] | 48.0 [39.71 to 56.29] | 42.0 [34.50 to 49.50] | 52.7 [36.62 to 68.72]
  Sweetness | 23.3 [8.96 to 37.71] | 25.8 [13.87 to 37.63] | 16.3 [7.09 to 25.41] | 23.9 [9.52 to 38.32]
  Sourness | 42.8 [27.34 to 58.16] | 29.3 [18.51 to 40.15] | 24.6 [13.38 to 35.79] | 18.8 [9.50 to 28.00]
  Saltiness | 34.6 [18.98 to 50.19] | 22.3 [11.42 to 33.24] | 21.1 [9.12 to 33.04] | 22.1 [11.27 to 32.89]
  Tongue/Mouth Burn | 23.4 [11.20 to 35.63] | 18.8 [8.54 to 28.96] | 15.8 [6.09 to 25.57] | 16.0 [5.18 to 26.82]
  Overall Liking | 70.7 [56.77 to 84.57] | 53.2 [40.38 to 65.96] | 42.5 [32.88 to 52.12] | 51.0 [34.37 to 67.63]

4. Primary Outcome: Mean Score of Sensory Attributes Based on Palatability Assessment Questionnaire at 20 Minutes Post-dose on Day 1
Description: as for outcome 1
Time Frame: At 20 minutes after tasting specified study formulation on Day 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Formulation A | Formulation B | Formulation C | Formulation D
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale
  Mouth Feel | 58.3 [45.28 to 71.39] | 41.5 [28.32 to 54.68] | 29.8 [20.42 to 39.08] | 44.5 [28.50 to 60.50]
  Bitterness | 62.7 [48.64 to 76.69] | 46.0 [35.17 to 56.83] | 24.0 [15.55 to 32.45] | 47.8 [31.64 to 64.03]
  Sweetness | 19.1 [7.53 to 30.64] | 26.6 [14.90 to 38.26] | 16.5 [8.20 to 24.80] | 22.0 [8.62 to 35.38]
  Sourness | 40.4 [25.64 to 55.19] | 26.3 [14.97 to 37.70] | 19.5 [8.98 to 30.02] | 26.3 [11.96 to 40.54]
  Saltiness | 33.8 [18.87 to 48.80] | 18.9 [9.03 to 28.80] | 18.8 [8.48 to 29.19] | 21.3 [9.04 to 33.63]
  Tongue/Mouth Burn | 23.5 [10.16 to 36.84] | 16.8 [7.33 to 26.17] | 14.8 [5.59 to 24.08] | 13.5 [4.11 to 22.89]
  Overall Liking | 69.4 [53.71 to 85.12] | 49.4 [36.99 to 61.85] | 34.7 [25.77 to 43.57] | 46.8 [29.96 to 63.71]

5. Primary Outcome: Mean Score of Sensory Attributes Based on Palatability Assessment Questionnaire at 1 Minute Post-dose on Day 2
Description: as for outcome 1
Time Frame: At 1 minute after tasting specified study formulation on Day 2
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Data was reported only for those formulations which were administered on Day 2.
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Groups:
- Formulation E: Participants received single dose of formulation E of sisunatovir. Participants had to swirl the formulation in the mouth for approximately 10 seconds, and then spit it out.
- Formulation F: Participants received single dose of formulation F of sisunatovir. Participants had to swirl the formulation in the mouth for approximately 10 seconds, and then spit it out.
Arm/Group | Formulation A | Formulation E | Formulation F
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale
  Mouth Feel | 61.6 [49.91 to 73.25] | 39.8 [29.68 to 49.99] | 46.7 [31.54 to 61.79]
  Bitterness | 61.8 [50.27 to 73.23] | 43.4 [33.09 to 53.74] | 48.3 [35.96 to 60.54]
  Sweetness | 24.8 [14.14 to 35.53] | 39.3 [29.25 to 49.25] | 38.3 [25.68 to 50.82]
  Sourness | 36.7 [25.23 to 48.11] | 27.0 [15.86 to 38.14] | 28.8 [16.81 to 40.86]
  Saltiness | 41.2 [27.39 to 54.94] | 21.9 [11.17 to 32.67] | 28.0 [16.41 to 39.59]
  Tongue/Mouth Burn | 22.8 [10.79 to 34.88] | 20.2 [8.80 to 31.54] | 20.1 [8.96 to 31.21]
  Overall Liking | 68.3 [56.89 to 79.61] | 42.7 [31.95 to 53.38] | 48.3 [32.68 to 63.99]

6. Primary Outcome: Mean Score of Sensory Attributes Based on Palatability Assessment Questionnaire at 5 Minutes Post-dose on Day 2
Description: as for outcome 1
Time Frame: At 5 minutes after tasting specified study formulation on Day 2
Population: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Formulation A | Formulation E | Formulation F
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale
  Mouth Feel | 53.3 [41.57 to 65.09] | 38.4 [24.10 to 52.74] | 42.3 [27.08 to 57.42]
  Bitterness | 61.2 [51.02 to 71.32] | 46.7 [31.81 to 61.52] | 48.7 [34.50 to 62.83]
  Sweetness | 21.7 [10.87 to 32.47] | 29.5 [17.59 to 41.41] | 32.8 [20.13 to 45.37]
  Sourness | 41.0 [30.06 to 51.94] | 26.8 [17.45 to 36.21] | 26.9 [17.27 to 36.56]
  Saltiness | 33.6 [19.72 to 47.44] | 22.3 [11.40 to 33.10] | 22.7 [10.99 to 34.35]
  Tongue/Mouth Burn | 20.3 [8.84 to 31.66] | 19.6 [8.36 to 30.80] | 19.7 [8.81 to 30.52]
  Overall Liking | 62.5 [50.35 to 74.65] | 43.0 [27.13 to 58.87] | 44.3 [28.48 to 60.18]

7. Primary Outcome: Mean Score of Sensory Attributes Based on Palatability Assessment Questionnaire at 10 Minutes Post-dose on Day 2
Description: as for outcome 1
Time Frame: At 10 minutes after tasting specified study formulation on Day 2
Population: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Formulation A | Formulation E | Formulation F
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale
  Mouth Feel | 52.5 [40.28 to 64.72] | 39.0 [24.59 to 53.41] | 38.2 [24.25 to 52.08]
  Bitterness | 56.9 [44.66 to 69.17] | 45.1 [31.67 to 58.50] | 42.7 [30.51 to 54.83]
  Sweetness | 20.1 [8.97 to 31.20] | 27.5 [14.74 to 40.26] | 31.3 [18.64 to 44.03]
  Sourness | 39.7 [27.79 to 51.54] | 29.3 [19.41 to 39.09] | 22.8 [12.36 to 33.30]
  Saltiness | 31.5 [18.02 to 44.98] | 20.4 [9.51 to 31.32] | 20.5 [9.38 to 31.62]
  Tongue/Mouth Burn | 20.8 [8.76 to 32.74] | 18.8 [7.92 to 29.58] | 19.0 [8.16 to 29.84]
  Overall Liking | 59.3 [45.12 to 73.38] | 43.2 [27.24 to 59.10] | 42.9 [26.72 to 59.11]

8. Primary Outcome: Mean Score of Sensory Attributes Based on Palatability Assessment Questionnaire at 20 Minutes Post-dose on Day 2
Description: as for outcome 1
Time Frame: At 20 minutes after tasting specified study formulation on Day 2
Population: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Formulation A | Formulation E | Formulation F
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale
  Mouth Feel | 48.9 [36.89 to 60.94] | 35.6 [21.51 to 49.65] | 37.1 [21.61 to 52.55]
  Bitterness | 54.2 [41.67 to 66.67] | 40.8 [27.43 to 54.24] | 43.0 [29.76 to 56.24]
  Sweetness | 19.2 [8.30 to 30.03] | 26.2 [12.80 to 39.53] | 27.4 [14.90 to 39.94]
  Sourness | 39.8 [27.45 to 52.05] | 25.3 [16.37 to 34.13] | 23.3 [12.91 to 33.75]
  Saltiness | 32.0 [18.83 to 45.17] | 20.2 [9.36 to 30.97] | 20.1 [9.73 to 30.43]
  Tongue/Mouth Burn | 19.6 [8.17 to 31.00] | 17.6 [7.08 to 28.08] | 18.1 [7.56 to 28.61]
  Overall Liking | 58.4 [43.08 to 73.76] | 42.1 [25.84 to 58.33] | 38.3 [21.04 to 55.62]

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE was an AE that occurred after initiation of study intervention (formulation) that was not present at the time of treatment start up to 35 days after administration of last study intervention (formulation).
Time Frame: Day 1 of receiving formulation up to 35 days after last formulation of the study (up to 37 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Formulation A | Formulation B | Formulation C | Formulation D | Formulation E | Formulation F
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
Participants | 0 | 3 | 0 | 0 | 1 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Laboratory analysis included were: hematology, chemistry and urinalysis. Clinically significance in laboratory abnormalities were judged by investigator.
Time Frame: 1 day prior to first formulation (Day -1) up to last formulation on Day 2 (up to 3 days)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Formulation A | Formulation B | Formulation C | Formulation D | Formulation E | Formulation F
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Vital signs included blood pressure (systolic and diastolic) and pulse rate. Clinically significance in vital sign abnormalities were judged by investigator.
Time Frame: Day 1 of receiving formulation up to last formulation on Day 2 (up to 2 days)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Formulation A | Formulation B | Formulation C | Formulation D | Formulation E | Formulation F
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of receiving formulation up to 35 days after last formulation of the study (up to 37 days)
Description: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Arm/Group | Formulation A | Formulation B | Formulation C | Formulation D | Formulation E | Formulation F
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 3/12 | 0/12 | 0/12 | 1/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Formulation A (N=12) | Formulation B (N=12) | Formulation C (N=12) | Formulation D (N=12) | Formulation E (N=12) | Formulation F (N=12)
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT06003829/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT06003829/SAP_001.pdf